CLINICAL TRIAL: NCT04330404
Title: Effects of Cognitive Strategy Training on Daily Function in People With Subjective Cognitive Decline
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Shu-Chen Liu, Graduate student, Department of Occupational Therapy, College of Medicine, National Cheng Kung University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCKU HREC-E-108-388-2
Record Dates: First submitted 2019-12-22; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Subjective Cognitive Decline

STUDY DESIGN:
Intervention Model Description: The experimental group will receive the Cognitive strategy training. The active control group will receive group interactive game.
Who Masked: Outcomes Assessor
Masking Description: For the interventionist, it is important to build relationships with participants through baseline interviews. The pre-test will be conducted by the interventionist. Assessors at post-intervention, and 3-month follow-up will be blind to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive strategy training (Experimental): The experimental group will receive the Cognitive strategy training (CST), which includes awareness enhancement, cognitive-related education, discussion of everyday cognitive difficulties, generation of cognitive strategies, cognitive strategy practice, and homework assignments.
  Interventions: Behavioral: Cognitive strategy training
- group interactive game (Active Comparator): The active control group will receive group interactive game, including table games and games using songs, balloons, newspapers and so on.
  Interventions: Behavioral: group interactive game

INTERVENTIONS:
Behavioral: Cognitive strategy training — The Cognitive strategy training, including awareness enhancement, cognitive-related education, discussion of everyday cognitive difficulties, generation of cognitive strategies, cognitive strategy practice, and homework assignments
  Arms: Cognitive strategy training
Behavioral: group interactive game — The active control group will receive group interactive game, including table games and games using songs, balloons, newspapers and so on.
  Arms: group interactive game

SUMMARY:
Subjective cognitive decline (SCD) is the transitional state between normal aging and mild cognitive impairment. SCD is defined as having self-perceived declines in any cognitive domain over time; having normal performance on cognitive testing; no dementia or depression. Cognitive difficulties can lead to a decline on daily function and quality of life. Early intervention can prevent SCD from developing into dementia.

Cognitive strategy training (CST) aims to generate individualized strategies to solve cognitive problems, which can be effective to improve daily functions and performances. However, there is limited clinical research aimed at improving daily functions for SCD. Most non-pharmacological studies have conducted objective cognitive training, which may not enhance daily performance. Previous studies also seldom examine the effectiveness of the intervention to improve daily function, quality of life, self-efficacy and motivation.

This study adopts a quasi-experimental design. The investigators will recruit 80 community-dwelling people with SCD who are aged 55 and older. There will be 40 participants in each group. The experimental group will receive the CST. The active control group will receive group interactive game. Both groups will have 8 sessions for one hour per week for a total of 8 weeks. Outcome measures include daily function, self-efficacy, motivation for change, and quality of life. Assessments will be performed at baseline, post-intervention, and 3-month follow-up. The demographic data of the two groups will be compared using the independent sample t-test and chi-square test. Changes on outcomes between the two groups will be analyzed by two-way ANOVA. This study was approved by the Human Research Ethics Committee at National Cheng Kung University. All participants provided written informed consent before testing.

This study aims to (1) examine the feasibility of the CST in community-dwelling people with SCD; (2) explore the efficacy of the CST on daily function, self-efficacy, motivation for change, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* aged 55 and above
* live in community
* self-perceived decline in cognition compared to five years ago
* subjective cognitive decline, Cognitive Failure Questionnaire (CFQ) score above zero.

Exclusion Criteria:

* objective cognitive impairment, Taiwanese version of the Montreal Cognitive Assessment (MoCA-T) scores below 24
* any medical, neurological or psychiatric disorders, Brief Symptom Rating Scale (BSRS-5) scores 10 or more
* severe visual, auditory, verbal or physical impairments interfere with communication, command compliance, and strategy execution
* participate in other research related to cognitive strategy at the same time.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Canadian Occupational Performance Measure-Chinese version (COPM-C) at post-intervention, and 3-month follow-up. | Assessments will be performed at baseline, within one week after the intervention, and 3-month follow-up after the intervention. .
  Canadian Occupational Performance Measure-Chinese version (COPM-C) is a semi-structured interview questionnaire used to assess self-perceived problems in occupational performance areas.
  Participants need to identify cognitive-related occupational performance problems, then score the importance from 1 to 10. The higher the score, the more important it is.
  Participants also need to score their performance and satisfaction from 1 to 10 on the first five important issues. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Change from Baseline General Self-Efficacy Scale (GSE) at post-intervention, and 3-month follow-up. | Assessments will be performed at baseline, within one week after the intervention, and 3-month follow-up after the intervention.
  General Self-Efficacy Scale (GSE) is a self-reported questionnaire used to assess individual beliefs of how effective they are in facing stress and challenges. The scale scores range from 10 to 40, with higher scores indicating better self-efficacy.
Change from Baseline Contemplation ladder at post-intervention, and 3-month follow-up. | Assessments will be performed at baseline, within one week after the intervention, and 3-month follow-up after the intervention.
  Contemplation ladder is an 11-point scale used to assess readiness and motivation for change before action. The scale score is between 0 and 10, with higher scores indicating greater motivation for change.
Change from Baseline COOP/WONCA (World Organization of Family Doctors) charts at post-intervention, and 3-month follow-up. | Assessments will be performed at baseline, within one week after the intervention, and 3-month follow-up after the intervention.
  COOP/WONCA (World Organization of Family Doctors) is a self-reported chart used to assess health-related quality of life. The scale scores range from 6 to 30, with lower scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Shuchen Liu, Principal Investigator — Department of Occupational Therapy, College of Medicine, National Cheng Kung University, Taiwan
Locations (1):
- Department of Occupational Therapy, College of Medicine, National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No